CLINICAL TRIAL: NCT01359644
Title: Parallel, Open-Label, Randomized Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of PSI-7977 in Combination With BMS-790052 With or Without Ribavirin in Treatment Naive Subjects Chronically Infected With Hepatitis C Virus Genotypes 1, 2, or 3
Brief Title: Study to Determine the Safety and Effectiveness of Antiviral Combination Therapy to Treat Hepatitis C Virus (HCV) in Patients Who Have Previously Not Received the Standard of Care
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pharmasset (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI444-040
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Results first posted 2015-10-23 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Sofosbuvir; daclatasvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Treatment A: PSI-7977 + Daclatasvir (Experimental): Genotype 1a or 1b
  Interventions: Drug: PSI-7977; Drug: Daclatasvir
- Treatment B: PSI-7977 + Daclatasvir (Experimental): Genotype 2 or 3
  Interventions: Drug: PSI-7977; Drug: Daclatasvir
- Treatment C: PSI-7977 + Daclatasvir (Experimental): Genotype 1a or 1b
  Interventions: Drug: PSI-7977; Drug: Daclatasvir
- Treatment D: PSI-7977 + Daclatasvir (Experimental): Genotype 2 or 3
  Interventions: Drug: PSI-7977; Drug: Daclatasvir
- Treatment E: PSI-7977 + Daclatasvir + Ribavirin (Experimental): Genotype 1a or 1b
  Interventions: Drug: PSI-7977; Drug: Daclatasvir; Drug: Ribavirin
- Treatment F: PSI-7977 + Daclatasvir+ Ribavirin (Experimental): Genotype 2 or 3
  Interventions: Drug: PSI-7977; Drug: Daclatasvir; Drug: Ribavirin
- Treatment G: PSI-7977 + Daclatasvir (Experimental): Hepatitis C virus genotype 1, treatment-naive patients
  Genotype 1a or 1b
  Interventions: Drug: PSI-7977; Drug: Daclatasvir
- Treatment H: PSI-7977 + BMS-790052 + Ribavirin (Experimental): Hepatitis C virus genotype 1, treatment-naive patients
  Genotype 1a or 1b
  Interventions: Drug: PSI-7977; Drug: Daclatasvir; Drug: Ribavirin
- Treatment I: PSI-7977 + Daclatasvir (Experimental): Patients who experienced telaprevir/boceprevir treatment failure
  Genotype 1a or 1b
  Interventions: Drug: PSI-7977; Drug: Daclatasvir
- Treatment J: PSI-7977 + Daclatasvir + Ribavirin (Experimental): Patients who experienced telaprevir/boceprevir treatment failure
  Genotype 1a or 1b
  Interventions: Drug: PSI-7977; Drug: Daclatasvir; Drug: Ribavirin

INTERVENTIONS:
Drug: PSI-7977 — Tablets, oral, 400 mg, once daily
Drug: Daclatasvir — Tablets, oral, 60 mg, once daily
  Other Names: BMS-790052
Drug: Ribavirin — Tablets, oral, 200 mg
  Other Names: Copegus ®
  Arms: Treatment E: PSI-7977 + Daclatasvir + Ribavirin; Treatment F: PSI-7977 + Daclatasvir+ Ribavirin; Treatment H: PSI-7977 + BMS-790052 + Ribavirin; Treatment J: PSI-7977 + Daclatasvir + Ribavirin

SUMMARY:
The purpose of the study is to determine whether therapy with the combination of PSI-7977 and daclatasvir (BMS-790052) with or without ribavirin is effective in treating hepatitis C virus (HCV) infection when given for 12 or 24 weeks as measured by sustained virologic response with undetectable HCV RNA 12 weeks post treatment

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18 to 70 years.
* Participants infected with hepatitis C virus (HCV) genotype 1, 2, or 3, with no previous exposure to an interferon formulation (ie, interferon-alpha, pegylated interferon-alpha) ribavirin, or other HCV-specific direct-acting antiviral (including daclatasvir and PSI-7977).
* Patients should have chronic hepatitis C genotype 1a, 1b, 2, or 3 as documented by: positive test results for anti-HCV antibody; HCV RNA; or a HCV genotype at least 6 months prior to screening, and HCV RNA and anti-HCV antibody at the time of screening.

Exclusion Criteria:

* Evidence of a medical condition associate with chronic liver disease other than HCV.
* History of variceal bleeding, hepatic encephalopathy, or ascites requiring management with diuretics or paracentesis.
* History of hemophilia.
* History of torsade de pointes.
* Current or known history of cancer (except in situ carcinoma of the cervix or adequately treated basal or squamous cell carcinoma of the skin) within 5 years prior to enrollment.
* History of gastrointestinal disease or surgical procedure (except cholecystectomy).
* History of clinically significant cardiac disease.
* Blood transfusion within 4 weeks prior to study drug administration.
* Poor venous access.
* Any other medical, psychiatric, and/or social reason which, in the opinion of the Investigator, would make the candidate inappropriate for participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (18):
- United States (17):
  - Southern California Liver Centers, Coronado, California
  - Research And Education, Inc., San Diego, California
  - University Of Colorado Denver & Hospital, Aurora, Colorado
  - University Of Florida Hepatology, Gainesville, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Miami Research Associates, South Miami, Florida
  - Mercy Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Lutherville, Maryland
  - University Of Michigan Health System, Ann Arbor, Michigan
  - Weill Cornell Medical College, New York, New York
  - Bronx Va Medical Center 3c Sub-J, The Bronx, New York
  - Options Health Research, Llc, Tulsa, Oklahoma
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - Alamo Medical Research, San Antonio, Texas
  - Metropolitan Research, Annandale, Virginia
  - Dean Clinic, Madison, Wisconsin
- Local Institution, San Juan, Puerto Rico

REFERENCES:
- [Derived] Sulkowski MS, Gardiner DF, Rodriguez-Torres M, Reddy KR, Hassanein T, Jacobson I, Lawitz E, Lok AS, Hinestrosa F, Thuluvath PJ, Schwartz H, Nelson DR, Everson GT, Eley T, Wind-Rotolo M, Huang SP, Gao M, Hernandez D, McPhee F, Sherman D, Hindes R, Symonds W, Pasquinelli C, Grasela DM; AI444040 Study Group. Daclatasvir plus sofosbuvir for previously treated or untreated chronic HCV infection. N Engl J Med. 2014 Jan 16;370(3):211-21. doi: 10.1056/NEJMoa1306218. PMID 24428467
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 18 centres in 2 countries.
Pre-assignment Details: A total of 350 participants were enrolled, and 211 were randomized and received study drug.
Groups:
- Treatment A: Sofosbuvir + Daclatasvir: Participants with hepatitis C virus (HCV) genotypes 1a or 1b received sofosbuvir, 400 mg, once daily for 7 days and then added daclatasvir, 60 mg, once daily for 24 weeks.
- Treatment B: Sofosbuvir + Daclatasvir: Participants with genotype 2 or 3 received sofosbuvir, 400 mg, once daily for 7 days and then added daclatasvir, 60 mg, once daily for 24 weeks.
- Treatment C: Sofosbuvir + Daclatasvir: Participants with genotype 1a or 1b received sofosbuvir, 400 mg, once daily and daclatasvir, 60 mg, once daily for 24 weeks.
- Treatment D: Sofosbuvir + Daclatasvir: Participants with genotype 2 or 3 received sofosbuvir, 400 mg, once daily and daclatasvir, 60 mg, once daily for 24 weeks.
- Treatment E: Sofosbuvir + Daclatasvir + Ribavirin: Participants with genotype 1a or 1b received sofosbuvir, 400 mg, once daily; daclatasvir, 60 mg, once daily for 24 weeks; and ribavirin in a total daily dose of 1000 mg (2 200-mg tablets AM and 3 200-mg tablets PM) for participants weighing <75 kg and a total daily dose of 1200 mg (3 200-mg tablets AM and 3 200-mg tablets PM) for participants weighing ≥75 kg for 24 weeks.
- Treatment F: Sofosbuvir + Daclatasvir + Ribavirin: Participants with genotype 2 or 3 received sofosbuvir, 400 mg, once daily; daclatasvir, 60 mg, once daily for 24 weeks; and ribavarin in total daily dose of 800 mg (2 200-mg tablets AM and 2 200-mg tablets PM) for 24 weeks.
- Treatment G: Sofosbuvir + Daclatasvir: Participants with genotype 1a or 1b received sofosbuvir, 400 mg, once daily and daclatasvir, 60 mg, once daily for 12 weeks.
- Treatment H : Sofosbuvir + Daclatasvir + Ribavirin: Participants with genotype 1a or 1b received sofosbuvir, 400 mg, once daily, daclatasvir, 60 mg, once daily for 12 weeks and ribavirin (in a total daily dose of 1000 mg (2 200-mg tablets AM and 3 200-mg tablets PM for participants weighing <75 kg and a total daily dose of 1200 mg (3 200-mg tablets AM and 3 200-mg tablets PM for participants weighing ≥ 75 kg) for 12 weeks.
- Treatment I: Sofosbuvir + Daclatasvir: Participants with genotype 1a or 1b who experienced telaprevir/boceprevir treatment failure received sofosbuvir, 400 mg, once daily and daclatasvir, 60 mg, once daily for 24 weeks.
- Treatment J: Sofosbuvir + Daclatasvir + Ribavirin: Participants with genotype 1a or 1b who experienced telaprevir/boceprevir treatment failure received sofosbuvir, 400 mg, once daily, daclatasvir, 60 mg, once daily for 24 weeks and ribavirin (in a total daily dose of 1000 mg (2 200-mg tablets AM and 3 200-mg tablets PM for participants weighing <75 kg and a total daily dose of 1200 mg (3 200-mg tablets AM and 3 200-mg tablets PM for participants weighing ≥75 kg) for 24 weeks.
Period: Treatment Period
Arm/Group | Treatment A: Sofosbuvir + Daclatasvir | Treatment B: Sofosbuvir + Daclatasvir | Treatment C: Sofosbuvir + Daclatasvir | Treatment D: Sofosbuvir + Daclatasvir | Treatment E: Sofosbuvir + Daclatasvir + Ribavirin | Treatment F: Sofosbuvir + Daclatasvir + Ribavirin | Treatment G: Sofosbuvir + Daclatasvir | Treatment H : Sofosbuvir + Daclatasvir + Ribavirin | Treatment I: Sofosbuvir + Daclatasvir | Treatment J: Sofosbuvir + Daclatasvir + Ribavirin
Started | 15 | 16 | 14 | 14 | 15 | 14 | 41 | 41 | 21 | 20
Completed | 15 | 15 | 13 | 14 | 15 | 12 | 41 | 41 | 21 | 20
Not Completed | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Follow-up Period
Arm/Group | Treatment A: Sofosbuvir + Daclatasvir | Treatment B: Sofosbuvir + Daclatasvir | Treatment C: Sofosbuvir + Daclatasvir | Treatment D: Sofosbuvir + Daclatasvir | Treatment E: Sofosbuvir + Daclatasvir + Ribavirin | Treatment F: Sofosbuvir + Daclatasvir + Ribavirin | Treatment G: Sofosbuvir + Daclatasvir | Treatment H : Sofosbuvir + Daclatasvir + Ribavirin | Treatment I: Sofosbuvir + Daclatasvir | Treatment J: Sofosbuvir + Daclatasvir + Ribavirin
Started | 15 | 16 | 14 | 14 | 15 | 13 | 41 | 41 | 21 | 20
Completed | 15 | 16 | 14 | 14 | 15 | 12 | 40 | 39 | 21 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment A: Sofosbuvir + Daclatasvir: Participants with hepatitis C virus genotype 1a or 1b received sofosbuvir, 400 mg, once daily for 7 days and then added daclatasvir, 60 mg, once daily for 24 weeks.
- Treatment: Sofosbuvir + Daclatasvir: Participants with genotype 2 or 3 received sofosbuvir, 400 mg, once daily for 7 days and then added daclatasvir, 60 mg, once daily for 24 weeks.
- Treatment D: Sofosbuvir + Daclatasvir: Participants with genotype-2 or -3 received sofosbuvir, 400 mg, once daily and daclatasvir, 60 mg, once daily for 24 weeks..
- Treatment E: Sofosbuvir +Daclatasvir + Ribavirin: Participants with genotype 1a or 1b received sofosbuvir, 400 mg, once daily; daclatasvir, 60 mg, once daily for 24 weeks; and ribavirin in a total daily dose of 1000 mg (2 200-mg tablets AM and 3 200-mg tablets PM) for participants weighing <75 kg and a total daily dose of 1200 mg (3 200-mg tablets AM and 3 200-mg tablets PM) for participants weighing ≥75 kg for 24 weeks.
- Treatment G: Sofosbuvir + Daclatasvir: Participants with genotype1 a or 1b received sofosbuvir, 400 mg, once daily and daclatasvir, 60 mg, once daily for 12 weeks..
- Treatment H: Sofosbuvir +Daclatasvir + Ribavirin: Participants with genotype 1a or 1b received sofosbuvir, 400 mg, once daily, daclatasvir, 60 mg, once daily for 12 weeks and ribavirin (in a total daily dose of 1000 mg (2 200-mg tablets AM and 3 200-mg tablets PM for participants weighing <75 kg and a total daily dose of 1200 mg (3 200-mg tablets AM and 3 200-mg tablets PM for participants weighing ≥ 75 kg) for 12 weeks.
- Treatment I: Sofosbuvir + Daclatasvir: Participants with genotype 1a or 1b who experienced telaprevir/boceprevir treatment failure received sofosbuvir, 400 mg once daily and daclatasvir, 60 mg, once daily for 24 weeks.
- Treatment J: Sofosbuvir +Daclatasvir +Ribavirin: Participants with genotype 1a or 1b who experienced telaprevir/boceprevir treatment failure received sofosbuvir, 400 mg once daily, daclatasvir, 60 mg, once daily for 24 weeks and ribavarin in a total daily dose of 1000 mg (2 200-mg tablets AM and 3 200-mg tablets PM for participants weighing <75 kg) and a total daily dose of 1200 mg (3 200-mg tablets AM and 3 200-mg tablets PM for participants weighing ≥75 kg) for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Treatment A: Sofosbuvir + Daclatasvir | Treatment: Sofosbuvir + Daclatasvir | Treatment C: Sofosbuvir + Daclatasvir | Treatment D: Sofosbuvir + Daclatasvir | Treatment E: Sofosbuvir +Daclatasvir + Ribavirin | Treatment F: Sofosbuvir + Daclatasvir + Ribavirin | Treatment G: Sofosbuvir + Daclatasvir | Treatment H: Sofosbuvir +Daclatasvir + Ribavirin | Treatment I: Sofosbuvir + Daclatasvir | Treatment J: Sofosbuvir +Daclatasvir +Ribavirin | Total
Number analyzed (Participants) | 15 | 16 | 14 | 14 | 15 | 14 | 41 | 41 | 21 | 20 | 211
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (10.18) | 50.6 (8.53) | 52.7 (7.39) | 49.7 (10.49) | 50.9 (11.72) | 48.8 (12.27) | 50.9 (11.56) | 53.1 (9.53) | 56.6 (9.89) | 52.6 (10.89) | 52.0 (10.37)
Age, Customized [Number; unit: participants]
  <65 years | 15 | 15 | 14 | 13 | 15 | 13 | 39 | 38 | 18 | 19 | 199
  >= 65 years | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 3 | 3 | 1 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 5 | 8 | 8 | 9 | 21 | 20 | 8 | 8 | 100
  Male | 7 | 11 | 9 | 6 | 7 | 5 | 20 | 21 | 13 | 12 | 111

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response at Post Treatment Week 12 (SVR12)
Description: SVR12 was defined as hepatitis C virus (HCV) RNA less than the lower limit of quantitation, target detected or target not detected (ie, HCV RNA <25 IU/mL) at follow-up Week 12. DCV=daclatasvir, SOF=sofosbuvir.
Time Frame: Follow-up Week 12
Population: The analysis was performed in all treated participants who received at least 1 dose of active study therapy. The 'n' signifies those participants evaluable for this measure at specified time points for each group, respectively.
Measure: Number; unit: Percentage of participants
Groups:
- Treatment-naive Participants With Genotype 1: Participants with genotype 1a or 1b and no previous exposure to an interferon formulation, ribavirin, or other hepatitis C virus-specific direct acting antiviral received sofosbuvir, 400 mg + daclatasvir, 60 mg, ± ribavirin (a total daily dose of 1000 mg/1200 mg) tablets once daily for 12 or 24 weeks.
- Treatment-naive Participants With Genotype 2 or 3: Participants with genotype 2 or 3 and no previous exposure to an interferon formulation, ribavirin, or other hepatitis C virus-specific direct-acting antiviral received sofosbuvir, 400 mg + daclatasvir, 60 mg ± ribavirin (a total daily dose of 1000 mg/1200 mg) once daily for 12 or 24 weeks.
- Telaprevir or Boceprevir Failures With Genotype 1: Participants with genotype 1a or 1b who experienced telaprevir or boceprevir treatment failure received sofosbuvir, 400 mg + daclatasvir, 60 mg, tablets ± ribavirin (a total daily dose of 1000 mg/1200 mg) tablets once daily for 24 weeks.
Arm/Group | Treatment-naive Participants With Genotype 1 | Treatment-naive Participants With Genotype 2 or 3 | Telaprevir or Boceprevir Failures With Genotype 1
Number analyzed (Participants) | 126 | 44 | 41
Percentage of participants
  DCV/SOF with ribavirin (n=56, 14, 20) | 96.4 | 85.7 | 95.0
  DCV/SOF without ribavirin (n=70, 30, 21) | 100.0 | 93.3 | 100.0
  DCF/SOF All | 98.4 | 90.9 | 97.6

2. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at Post Treatment Week 24 (SVR24)
Description: SVR24 was defined as participant's hepatitis C virus RNA less than the lower limit of quantitation, target detected or target not detected at follow-up Week 24. DCV=daclatasvir, SOF=sofosbuvir.
Time Frame: Follow-up Week 24
Population: The analysis was performed in all treated participants who received at least 1 dose of active study therapy. Here the 'n' signifies those participants evaluable for this measure at specified time points for each group, respectively.
Measure: Number; unit: Percentage of participants
Groups:
- Treatment-naive Participants With Genotype 1: Participants with genotype 1a or 1b and no previous exposure to an interferon formulation or ribavirin or other hepatitis C virus-specific direct-acting antiviral received sofosbuvir 400 mg tablets + daclatasvir 60 mg tablets ± ribavirin (a total daily dose of 1000 mg/1200mg) tablets once daily for 12 or 24 weeks.
- Treatment-naive Participants With Genotype 2 or 3: Participants with genotype 2 or 3 and no previous exposure to an interferon formulation or ribavirin or other hepatitis C virus-specific direct-acting antiviral received sofosbuvir, 400 mg + daclatasvir, 60 mg ± ribavirin (a total daily dose of 1000 mg/1200 mg) once daily for 12 or 24 weeks.
- Telaprevir/Boceprevir Failures With Genotype 1: Participants with genotype 1a or 1b who experienced telaprevir or boceprevir treatment failure received sofosbuvir, 400 mg + daclatasvir, 60 mg, tablets ± ribavirin (a total daily dose of 1000 mg/1200 mg) tablets once daily for 24 weeks.
Arm/Group | Treatment-naive Participants With Genotype 1 | Treatment-naive Participants With Genotype 2 or 3 | Telaprevir/Boceprevir Failures With Genotype 1
Number analyzed (Participants) | 126 | 44 | 41
Percentage of participants
  DCV/SOF with ribavirin (n=56, 14, 20) | 94.6 | 92.9 | 100.0
  DCV/SOF without ribavirin (n=70, 30, 21) | 95.7 | 93.3 | 100.0
  DCV/SOF All | 95.2 | 93.2 | 100.0

3. Secondary Outcome: Percentage of Participants With Viral Breakthrough During the Treatment Period
Description: Viral breakthrough is defined as any confirmed increase in viral load ≥1 log from nadir or any confirmed hepatitis C virus RNA levels ≥25 IU/mL on or after Week 8.
Time Frame: First dose of study drug (Day 1) up to end of treatment period (up to 12 or 24 weeks, depending on treatment group)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Groups:
- Telaprevir or Boceprevir Failures With Genotype 1: Participants with genotype 1a or 1b who experienced telaprevir or boceprevir treatment failure received sofosbuvir, 400 mg + daclatasvir, 60 mg, tablets ± ribavirin (a total daily dose of 1000 mg/1200 mg) tablets once daily for 12 or 24 weeks.
Arm/Group | Treatment-naive Participants With Genotype 1 | Treatment-naive Participants With Genotype 2 or 3 | Telaprevir or Boceprevir Failures With Genotype 1
Number analyzed (Participants) | 126 | 44 | 41
Percentage of participants
  DCV/SOF with ribavirin (n=56, 14, 20) | 0 | 0 | 0
  DCV/SOF without ribavirin (n=70, 30, 21) | 0 | 3.3 | 0

4. Secondary Outcome: Percentage of Participants Who Experienced Viral Relapse During Follow-up Period
Description: Viral relapse during follow-up is defined as any confirmed quantifiable hepatitis C virus (HCV) RNA ≥25 IU/mL with HCV RNA levels less than the lower limit of quantitation, target detected or target not detected, ie, HCV RNA <25 IU/mL at the end of treatment.
Time Frame: Day 1 of follow-up period (Week 13 or 25, depending on treatment group) to end of follow-up period (up to 48 weeks)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment-naive Participants With Genotype 1 | Treatment-naive Participants With Genotype 2 or 3 | Telaprevir or Boceprevir Failures With Genotype 1
Number analyzed (Participants) | 126 | 44 | 41
Percentage of participants
  DCV/SOF with ribavirin (n=56, 14, 20) | 0 | 0 | 0
  DCV/SOF without ribavirin (n=70, 30, 21) | 1.4 | 3.3 | 0

5. Secondary Outcome: Change From Baseline in log10 Hepatitis C Virus (HCV) RNA at Follow-up Week 24
Description: Change from baseline in log10 HCV RNA at scheduled sampling time.
Time Frame: Baseline, Follow-up week 24
Population: The analysis was performed in all treated participants who received at least 1 dose of active study therapy.
Measure: Mean (Standard Deviation); unit: IU/mL
Groups:
- Treatment A: Sofosbuvir + Daclatasvir: Participants with hepatitis C virus genotypes 1a or 1b received sofosbuvir, 400 mg, once daily) for 7 days and then added daclatasvir, 60 mg, once daily for 24 weeks.
- Treatment D: Sofosbuvir + Daclatasvir: Participants with genotype 2 or 3 received with sofosbuvir, 400 mg, once daily, and daclatasvir, 60 mg, once daily for 24 weeks.
- Treatment H: Sofosbuvir + Daclatasvir + Ribavirin: Participants with genotype 1a or 1b received with sofosbuvir, 400 mg, once daily, daclatasvir, 60 mg, once daily for 12 weeks and ribavirin (a total daily dose of 1000 mg (2 200-mg tablets AM and 3 200-mg tablets) PM for participants weighing <75 kg and a total daily dose of 1200 mg (3 200-mg tablets AM and 3 200-mg tablets) PM for participants weighing ≥75 kg) for 12 weeks.
- Treatment I: Sofosbuvir + Daclatasvir: Participants with genotype 1a or 1b who experienced telaprevir/boceprevir treatment failure were administered with sofosbuvir, 400 mg, once daily, and daclatasvir, 60 mg, once daily for 24 weeks.
- Treatment J: Sofosbuvir + Daclatasvir + Ribavirin: Participants with genotype 1a or 1b who experienced telaprevir/boceprevir treatment failure received sofosbuvir, 400 mg, once daily; daclatasvir, 60 mg, once daily for 24 weeks; and ribavirin in a total daily dose of 1000 mg (2 200-mg tablets AM and 3 200-mg tablets PM) for participants weighing <75 kg and a total daily dose of 1200 mg (3 200-mg tablets at AM and 3 200-mg tablets PM) for participants weighing ≥75 kg for 24 weeks.
Arm/Group | Treatment A: Sofosbuvir + Daclatasvir | Treatment B: Sofosbuvir + Daclatasvir | Treatment C: Sofosbuvir + Daclatasvir | Treatment D: Sofosbuvir + Daclatasvir | Treatment E: Sofosbuvir + Daclatasvir + Ribavirin | Treatment F: Sofosbuvir + Daclatasvir + Ribavirin | Treatment G: Sofosbuvir + Daclatasvir | Treatment H: Sofosbuvir + Daclatasvir + Ribavirin | Treatment I: Sofosbuvir + Daclatasvir | Treatment J: Sofosbuvir + Daclatasvir + Ribavirin
Number analyzed (Participants) | 15 | 15 | 14 | 14 | 15 | 13 | 39 | 38 | 21 | 20
IU/mL
  Baseline | 1.28 (1.258) | 0.95 (0.0) | 0.95 (0.0) | 0.98 (0.114) | 0.95 (0.0) | 0.95 (0.0) | 0.95 (0.0) | 0.95 (0.0) | 0.95 (0.0) | 0.95 (0.0)
  Change at Follow-up week 24 | -5.19 (1.478) | -5.23 (1.601) | -5.67 (0.336) | -5.83 (0.509) | -5.77 (0.583) | -5.61 (0.610) | -5.19 (0.490) | -5.48 (0.576) | -5.39 (0.386) | -5.36 (0.380)

6. Secondary Outcome: Number of Participants Who Died and With Serious Adverse Events (SAEs) and Grade 3-4 Adverse Events (AEs), During the Treatment Period Prior to Addition of Rescue Therapy
Description: AE was defined as any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship with treatment. SAE was defined as a medical event that at any dose resulted in death, persistent or significant disability/incapacity, or drug dependency/abuse; was life-threatening, an important medical event, or a congenital anomaly/birth defect; or required or prolonged hospitalization. Based on the severity, AEs were categorized as Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4=Very severe.
Time Frame: First dose of study drug (Day 1) up to the start of rescue therapy (12 or 24 weeks, depending on treatment group)
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Groups:
- Daclatasvir + Sofosbuvir + Ribivirin (12 Weeks): Participants received sofosbuvir, 400 mg, once daily, daclatasvir, 60 mg, once daily for 12 weeks and ribavirin (a total daily dose of 1000 mg (2 200-mg tablets AM and 3 200-mg tablets) PM for participants weighing <75 kg and a total daily dose of 1200 mg (3 200-mg tablets AM and 3 200-mg tablets) PM for participants weighing ≥75 kg) for 12 weeks.
- Daclatasvir + Sofosbuvir With Ribivirin (24 Weeks): Participants received sofosbuvir, 400 mg, once daily, daclatasvir, 60 mg, once daily for 12 weeks and ribavirin (a total daily dose of 1000 mg (2 200-mg tablets AM and 3 200-mg tablets) PM for participants weighing <75 kg and a total daily dose of 1200 mg (3 200-mg tablets AM and 3 200-mg tablets) PM for participants weighing ≥75 kg) for 24 weeks.
- Daclatasvir + Sofosbuvir Without Ribivirin (12 Weeks); Daclatasvir + Sofosbuvir Without Ribivirin (24 Weeks): Participants received sofosbuvir, 400 mg, once daily, and daclatasvir, 60 mg, once daily for 12 weeks.
Arm/Group | Daclatasvir + Sofosbuvir + Ribivirin (12 Weeks) | Daclatasvir + Sofosbuvir With Ribivirin (24 Weeks) | Daclatasvir + Sofosbuvir Without Ribivirin (12 Weeks) | Daclatasvir + Sofosbuvir Without Ribivirin (24 Weeks)
Number analyzed (Participants) | 41 | 49 | 41 | 80
Participants
  Deaths | 0 | 0 | 0 | 0
  SAEs | 1 | 6 | 1 | 7
  AEs leading to discontinuation | 0 | 1 | 0 | 1
  Gr 3 Phosporus | 3 | 1 | 0 | 1
  Gr 3 Fasting serum glucose | 0 | 1 | 1 | 2
  Gr 3 Serum glucose | 0 | 2 | 0 | 1
  Gr 3 Total cholesterol | 1 | 0 | 0 | 1
  Gr 3 Uric acid | 1 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants Who Died and With Serious Adverse Events (SAEs), Grade 3-4 Adverse Events (AEs), and Grade 3-4 Abnormalities on Laboratory Test Results During Follow-up Period
Description: as for outcome 6
Time Frame: AEs: From Day 1 of follow-up period (Week 13 or 25) up to study discharge (up to 72 weeks). SAEs: From Day 1 of follow-up period (Week 13 or 25) up to 30 days after study discharge (up to 74 weeks)
Population: All participants who received at least 1 dose of study drug and entered follow-up period
Measure: Number; unit: Participants
Arm/Group | Daclatasvir + Sofosbuvir + Ribivirin (12 Weeks) | Daclatasvir + Sofosbuvir With Ribivirin (24 Weeks) | Daclatasvir + Sofosbuvir Without Ribivirin (12 Weeks) | Daclatasvir + Sofosbuvir Without Ribivirin (24 Weeks)
Number analyzed (Participants) | 41 | 48 | 41 | 80
Participants
  Deaths | 0 | 0 | 0 | 0
  SAEs | 2 | 4 | 2 | 4
  Grade 3-4 Lab Abnormalities: Serum glucose | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Treatment A: Sofosbuvir + Daclatasvir | Treatment B: Sofosbuvir + Daclatasvir | Treatment C: Sofosbuvir + Daclatasvir | Treatment D: Sofosbuvir + Daclatasvir | Treatment E: Sofosbuvir + Daclatasvir + Ribavirin | Treatment F: Sofosbuvir + Daclatasvir + Ribavirin | Treatment G: Sofosbuvir + Daclatasvir | Treatment H : Sofosbuvir + Daclatasvir + Ribavirin | Treatment I: Sofosbuvir + Daclatasvir | Treatment J: Sofosbuvir + Daclatasvir + Ribavirin
Serious Adverse Events (participants affected / at risk) | 2/15 | 0/16 | 2/14 | 3/14 | 2/15 | 2/14 | 1/41 | 1/41 | 0/21 | 2/20
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/14 | 0/14 | 0/15 | 0/14 | 0/41 | 0/41 | 0/21 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Sofosbuvir + Daclatasvir (N=15) | Treatment B: Sofosbuvir + Daclatasvir (N=16) | Treatment C: Sofosbuvir + Daclatasvir (N=14) | Treatment D: Sofosbuvir + Daclatasvir (N=14) | Treatment E: Sofosbuvir + Daclatasvir + Ribavirin (N=15) | Treatment F: Sofosbuvir + Daclatasvir + Ribavirin (N=14) | Treatment G: Sofosbuvir + Daclatasvir (N=41) | Treatment H : Sofosbuvir + Daclatasvir + Ribavirin (N=41) | Treatment I: Sofosbuvir + Daclatasvir (N=21) | Treatment J: Sofosbuvir + Daclatasvir + Ribavirin (N=20)
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suprapubic pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.